CLINICAL TRIAL: NCT06500910
Title: Exercise in Prematurely Born Preadolescents to Mitigate Cardiovascular Risk and Improve Cognitive Impairment
Acronym: EXCELSIOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henner Hanssen (Other)
Responsible Party: Sponsor-Investigator, Henner Hanssen, Professor, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-02358
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Training (Experimental): 10 weeks of exercise training
  Interventions: Other: Physical Exercise
- Control Group (No Intervention): Control group receiving age appropriate physical activity and life style recommendations as of current guidelines.

INTERVENTIONS:
Other: Physical Exercise — 10 weeks of child-friendly physical exercise program
  Other Names: Sports
  Arms: Exercise Training

SUMMARY:
EXCELSIOR is a randomized controlled trial to investigate the effect of physical exercise on cardiovascular health in prematurely born children. Participants will be randomly allocated to either an intervention group or a control group. The intervention will receive a child-friendly physical exercise program and the control group will receive age appropriate lifestyle- and exercise recommendations.

DETAILED DESCRIPTION:
Premature birth, i.e. the birth of babies before the 37th week of pregnancy, is an increasing challenge. Since the 1980s, medical advances such as special medication and ventilation techniques have significantly improved the chances of survival for premature babies. Worldwide, around 11% of all births are premature. Prematurity increases the risk of cardiovascular disease. Studies show that very premature babies have a significantly higher risk of heart problems. However, only little is known whether physical exercise could improve cardiovascular and cognitive function in prematurely born children.

All participants will undergo a baseline visit to assess vascular, cognitive and cardiopulmonary function. At the end of the visit, participants will be randomly allocated to either an intervention group or a control group. The intervention will receive a child-friendly physical exercise program and the control group will receive age appropriate lifestyle- and exercise recommendations. The physical exercise program is held 2-3 times per week for ten weeks targeting cardiovascular health and coordination. After 10 weeks, all participants will undergo a follow-up visit at which all measures will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls born prematurely (<= 32th week of gestation)
* aged 6 to 12 years
* informed consent provided

Exclusion Criteria:

* attendance of special education services related to attention disorders
* colour blindness or any chronic eye disorder
* being under pharmacological treatment for any mental disorder
* injuries, significant motor- or other disabilities which prohibit the participation in physical exercise
* visually provoked epilepsy
* children for whom no informed consent is provided

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-08-12 (Estimated); Study Completion 2025-08-12 (Estimated)

PRIMARY OUTCOMES:
Central Retinal Arteriolar Equivalent (CRAE) | 10 weeks
  Diameter of the retinal arterioles

CONTACTS AND LOCATIONS:
Overall Officials: Holger Burchert, PhD, Principal Investigator — University of Basel
Locations (1):
- Bereich Sport- und Bewegungsmedizin, Abteilung Präventive Sportmedizin & Systemphysiologie, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No